CLINICAL TRIAL: NCT02197715
Title: Improving Women's Sexual Health While in Drug Addiction Treatment
Brief Title: Sex and Female Empowerment
Acronym: SAFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-3075; R34DA033442 (NIH)
Record Dates: First submitted 2014-07-21; First posted 2014-07-23 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Opioid Use Disorder
Keywords: Pregnancy; Contraceptive Methods; Family Planning Services
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- computer-adaptive SAFE (Experimental): Computer-adaptive SAFE will consist of 4 60-minute sessions. Sessions 1 and 2 will explore participants' reasons to become and rewards for becoming pregnant/having children or avoiding it, introduce reproductive biology in the context of different contraceptive methods and explore the participant's ambivalence toward using different contraceptive methods. Session 3 will provide in-depth coverage of contraceptive methods and the need for use of a barrier method. Session 4 will focus on effective strategies to communicate with a sexual partner. Computer-adaptive SAFE will use an audio computer-assisted self-interviewing (ACASI) format.
  Interventions: Behavioral: Computer-adaptive SAFE
- Face-to-face SAFE (Experimental): Face-to-face SAFE will consist of 4 60-minute sessions using motivational interviewing techniques. Each session will be led by an experienced counselor. Sessions 1 and 2 will explore participants' reasons to become and rewards for becoming pregnant/having children or avoiding it, introduce reproductive biology in the context of different contraceptive methods and explore the participant's ambivalence toward using different contraceptive methods. Session 3 will provide in-depth coverage of contraceptive methods and the need for use of a barrier method, and relevant skills regarding how to use and negotiate use of contraceptive methods. Session 4 will focus on effective strategies to communicate with a sexual partner.
  Interventions: Behavioral: Face-to-face SAFE
- Usual Care (Active Comparator): Usual care comprises four 60-minute provider-led individual care sessions about HIV, STIs, and their risks, as well as prevention methods. Contraceptive methods are discussed within this context. There will be no demand on participants to attend these sessions. Participants will receive written take-home materials to review on their own and/or with their sex partners.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Computer-adaptive SAFE
  Arms: computer-adaptive SAFE
Behavioral: Face-to-face SAFE
  Arms: Face-to-face SAFE
Behavioral: Usual Care
  Arms: Usual Care

SUMMARY:
This study will develop and initially evaluate Sex and Female Empowerment (SAFE), an intervention designed to increase acceptance of and adherence to contraceptive practices among opioid-agonist-maintained women of childbearing age. The intervention will be delivered in one of two formats: a face-to-face brief intervention approach or a novel computer-adaptive platform. To the extent that either version of SAFE is found to be efficacious compared with usual care, it has the potential to reduce the number of unintended pregnancies and consequently decrease the need for and the costs of child protective services.

ELIGIBILITY:
Inclusion criteria will be:

1. ages 18-40 years old for women;
2. able to provide informed consent;
3. currently enrolled in a opioid-agonist-maintenance program;
4. currently not pregnant (urine testing confirmation);
5. report heterosexual orientation;
6. no tubal ligation or other sterilization;
7. no plans to become pregnant in the next 6 months; and
8. provides verifiable locator information.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Intervention Satisfaction | The earlier of the completion of the 4 interventions sessions or 6 weeks.
  Summary scale score: Derived from responses to a four-item 5-point Likert-type scale (1 = "not at all help" to 5 = "extremely helpful") of satisfaction with the intervention, administered at the end of each of the four intervention sessions.
Contraceptive Consultation Appointment | The earlier of the completion of the 4 intervention sessions or 6 weeks.
  Binary variable: Did or did not the participant schedule and attend an appointment with a obstetrical provider at University of North Carolina at Chapel Hill Obstetrical/Gynecological Services, determined from medical records.
Intervention Completion | The earlier of the completion of the 4 interventions sessions or 6 weeks.
  Binary variable: Completes or fails to complete all four intervention sessions in a 6-week period, determined from study records.
Contraceptive Method Effectiveness | The earlier of the completion of the 4 intervention sessions or 6 weeks.
  Percentage: The typical use effectiveness level of the contraceptive method in use at the end of the intervention based on responses to the National Survey of Family Growth contraceptive methods items. If the participant does not make an appointment and choose a contraceptive method, the typical-use effectiveness level of the contraceptive method indicated at intake in response to the Survey of Family Growth contraceptive methods items will be used. Typical effectiveness rating of contraceptive methods is a percentage between 15% and 99.85%, and will be based on Hatcher, R.A., Contraceptive technology, which reports success and failure rates for contraceptive methods in current use.

SECONDARY OUTCOMES:
Knowledge of Reproduction | Baseline, 1-, 3-, and 6-months post-baseline
  Summary scale score: Derived from eight true-false questions about participants' understanding of the information that was presented in the four intervention sessions about anatomy, menstruation, fertility, and conception, administered at each assessment time point.
Knowledge of Contraceptive Methods | Baseline, 1-, 3-, 6-months post-baseline
  Summary scale score: Derived from twenty true-false questions about participants' understanding of the information presented in the four intervention sessions about contraceptive methods, how hormonal contraceptives work, how to correctly use them; hormonal contraceptive side effects and ways to deal with them; which methods are effective against STIs/HIV; correct condom use, administered at each assessment time point.
Contraceptive Self-efficacy Scale | Baseline, 1-, 3-, and 6-months post-baseline
  Summary scale score: Derived from the Contraceptive Self-efficacy Scale, an eighteen-item 5-point Likert-type scale (1 = "not at all true of me" and 5 = "completely true of me") designed to measure a female respondent's motivational barriers to effective contraceptive use, including obtaining contraceptives, using contraceptives with a partner, talking to a partner about contraceptive use, using contraceptives despite partner approval, and preventing unprotected sexual intercourse, administered at each assessment time point.
Effective Contraceptive Behavior | Baseline, 1-, 3-, and 6-months post-baseline
  Ordered polytomous variable: Participant's self-report of their contraceptive behavior obtained at each assessment time point will be classified into 1 of 4 patterns: (1) "uninterrupted effective user" (e.g., implant, injectable, an IUD); (2) "uninterrupted other user" (use of effective methods on an interrupted basis); (3) "sporadic user" (use of some method when at risk for pregnancy); or (4) "nonuser", where "uninterrupted" in (1) means that an effective method was used for the entire time period under assessment; otherwise, categorized as (2).
Frequency of Use of Barrier Protection in past 30 days | Baseline, 1-, 3-, and 6-months post-baseline
  Count variable: Self-reported number of times in the past 30 days a participant used a barrier method for protection from HIV/STIs when engaging in sexual activities, collected at each assessment time point.
Number of Times Engaged in Unprotected Sex in past 30 days | Baseline, 1-, 3-, and 6-months post-baseline
  Count variable: Self-reported number of times in the past 30 days a participant engaged in unprotected vaginal, oral, or anal sex, collected at each assessment time point.

CONTACTS AND LOCATIONS:
Overall Officials: Hendrée E Jones, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Horizons, Chapel Hill, North Carolina, United States